CLINICAL TRIAL: NCT05907785
Title: Identification and Validation of Integrative Biomarkers of Physical Activity Level and Health in Children and Adolescents
Brief Title: Biomarkers of Physical Activity/health in Children and Adolescents
Acronym: INTEGRActiv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Fundación de Investigación Hospital General Universitario de Valencia (Unknown); Czech Academy of Sciences (Other); Aix Marseille Université (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INTEGRActiv; AC21_2/00033 (Other Grant/Funding Number: Instituto de Salud Carlos III - JPI HDHL)
Record Dates: First submitted 2023-05-05; First posted 2023-06-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-04

CONDITIONS: Physical Activity
Keywords: Integration analysis; Cardiorespiratory fitness; Metabolomics; Transcriptomics; miRNome; Adipokines; Cytokines; Biomarkers
MeSH Terms: conditions — Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: An educational intervention to improve physical activity and promote healthy dietary habits will be carried out in two groups of children/adolescents: (1) a prepubertal group and (2) a postpubertal group. Within each group, there will be volunteers with normal weight (NW), overweight (OW), and obesity (OB).
  A total of 180 volunteers will be assessed for eligibility (90 for each group), and 60 of them (30 for each group) will be allocated to study (intervention study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prepubertal group: Educational intervention (Experimental): An educational intervention to improve physical activity and promote healthy dietary habits will be carried out in prepubertal (8-10 years) volunteers with normal weight (NW), overweight (OW), and obesity (OB).
  Interventions: Behavioral: Educational intervention
- Postpubertal group: Educational intervention (Experimental): An educational intervention to improve physical activity and promote healthy dietary habits will be carried out in postpubertal (13-15 years) volunteers with normal weight (NW), overweight (OW), and obesity (OB).
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — The intervention will consist of recommendations to improve physical activity (PA) and dietary habits. It is based on the PAIDO Programme (www.programapaido.es), an outpatient family-based multidisciplinary programme that combines PA, education on nutrition, and behavioural therapy. It will last 6 months and improvement of metabolic health and body weight loss is expected, particularly in the groups with overweight and obesity. The dietary intervention will be focused on the promotion of the Mediterranean diet, with follow-up and advice from a dietitian-nutritionist. Participants will be encouraged in reducing sedentary behaviour (watching television, playing computer games, playing board games). Performance of aerobic and strength physical exercises will be scheduled, progressively increasing the intensity. Volunteers and their parents will participate in monthly sessions to follow-up on adherence to the PA and dietary recommendations and give personalized advice.

SUMMARY:
This clinical trial is aimed to recruit a core cohort of children and adolescents, and to perform an educational intervention and follow-up study in a subgroup of volunteers from this core cohort, to obtain specific measurements and samples of interest in these volunteers that will be used for identification and validation of the biomarkers of physical activity (PA) and health.

DETAILED DESCRIPTION:
Physical activity (PA) provides health benefits across the lifespan and improves many established cardiovascular risk factors that have a significant impact on overall mortality. Childhood and adolescence are critical periods for life-time health; processes underlying cardiovascular diseases and obesity generally originate in early ages. However, it is not clear how PA links to different parameters of health.

There is an important need to cover this critical gap and, more specifically, to have biomarkers allowing to relate the degree of PA with effects on health. INTEGRActiv addresses this new scientific and societal challenge by focusing on the identification of integrated markers reflecting both aspects - PA level and health - in children and adolescents, which represent an important target population to address personalized interventions to improve future, life long, metabolic health. Identification of new biomarkers will be achieved by combining measures of PA and cardiorespiratory and muscular fitness with anthropometric measures, cardiovascular risk factors and endocrine markers, cytokines, circulating miRNA, and gene expression profile in blood cells and metabolomics profile in plasma and blood cells.

Following identification in a core cohort and data integration analysis, candidate biomarkers will be further assessed in core cohort subjects after educational intervention and in existing samples from other independent studies. INTEGRActiv encompasses relevant progress beyond the state-of-the-art for a) the definition of potential biomarkers for PA level in childhood and adolescence; b) the provision of relevant mechanistic information for the link between PA and metabolic health in youth subjects; c) the identification of factors such as age, gender, body weight, sleep behavior and puberal status that quantitatively affect biomarker responses; d) the use and development of new tools in biomarker research, including integrative analysis; e) further assessment and first-step validation of promising candidate biomarkers in an intervention study and other independent studies. It is expected that new identified robust biomarkers reflecting PA level and its relation with health will guide nutritional/life-style and clinical advice and public policies related to endorse biomarker- based personalised PA, with a better adherence and response, to promote health and prevent disease risk factors since early stages of life.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian children/adolescents with age between 8-10 years for the prepubertal and 13-15 years for the postpubertal groups
* BMI z-score between those established by the World Health Organization for the subgroups with NW, OW or OB

Exclusion Criteria:

* Children/adolescents with reported pathologies
* Clinical recommendations against performance of physical activity
* Presence of eating disorders

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
BMI Z-score | Baseline (all groups)
  BMI z-score will be calculated from height and weight data, considering age and sex, following World Health Organization (WHO) guidelines.
BMI Z-score | 3 months (all groups)
  BMI z-score will be calculated from height and weight data, considering age and sex, following WHO guidelines.
BMI Z-score | 6 months (all groups)
  BMI z-score will be calculated from height and weight data, considering age and sex, following WHO guidelines.

SECONDARY OUTCOMES:
Weight | Baseline (all groups)
  Weight (kg)
Weight | 3 months (all groups)
  Weight (kg)
Weight | 6 months (all groups)
  Weight (kg)
Height | Baseline (all groups)
  Height (m)
Height | 3 months (all groups)
  Height (m)
Height | 6 months (all groups)
  Height (m)
Waist circumference | Baseline (all groups)
  Waist circumference (cm)
Waist circumference | 3 months (all groups)
  Waist circumference (cm)
Waist circumference | 6 months (all groups)
  Waist circumference (cm)
Body composition | Baseline (all groups)
  Lean and fat mass (in %) measured using bioimpedance
Body composition | 3 months (all groups)
  Lean and fat mass (in %) measured using bioimpedance
Body composition | 6 months (all groups)
  Lean and fat mass (in %) measured using bioimpedance
Blood pressure | Baseline (all groups)
  Systolic and diastolic pressure will be measured (mm Hg)
Blood pressure | 3 months (all groups)
  Systolic and diastolic pressure will be measured (mm Hg)
Blood pressure | 6 months (all groups)
  Systolic and diastolic pressure will be measured (mm Hg)
Handgrip strength | Baseline (all groups)
  Handgrip strength from right and left hands (Kg). This measure will be used, together with standing broad jump tests to assess musculoskeletal fitness.
Standing long jump | Baseline (all groups)
  Standing long jump (cm). This measure will be used, together with handgrip strenght to assess musculoskeletal fitness.
Cardiorespiratory Fitness (CRF) | Baseline (all groups)
  CRF will be measured as maximal oxygen consumption (V̇O2max) from cardiopulmonary exercise testing, using a treadmill test and the Balke protocol
Change in the level of physical activity (PA) during 6 months evaluated by accelerometry | Change from baseline in physical activity at 6 months (all groups)
  Different intensities of PA will be measured during one week before (baselline) and after the intervention (6 months) using accelerometry (actigraph GTX3+)
Adherence to the Mediterranean diet | Baseline (all groups)
  Adherence to the Mediterranean diet will be evaluated using the KIDMED, Mediterranean Diet Quality Index in children and adolescents. Score: 0-12. Value of the KIDMED score: ≤3, very-low-quality diet; 4-7, need to improve the food pattern to adjust it to the Mediterranean one; ≥8, optimal Mediterranean diet.
Adherence to the Mediterranean diet | 6 months (all groups)
  Adherence to the Mediterranean diet will be evaluated using the KIDMED, Mediterranean Diet Quality Index in children and adolescents. Score: 0-12. Value of the KIDMED score: ≤3, very-low-quality diet; 4-7, need to improve the food pattern to adjust it to the Mediterranean one; ≥8, optimal Mediterranean diet.
Physical activity (PA) level | Baseline (all groups)
  PA level will be evaluated using the Questionnaire for Older Children (PAQ-C) and for Adolescents (PAQ-A); score: 0-5 for different levels of PA (no units).
Physical activity (PA) level | 6 months (all groups)
  PA level will be evaluated using the Questionnaire for Older Children (PAQ-C) and for Adolescents (PAQ-A); score: 0-5 for different levels of PA (no units).
Sedentary behaviour | Baseline (all groups)
  Sedentary behaviour will be evaluated using a Screen Time Questionnaire (STQ). The total screen hours will ba obtained by measuring: hours of daily TV, weekend TV, daily Computer, weekend computer, daily videogames, weekend videogames, daily free internet, weekend free internet, daily study internet, weekend study internet, and weekend study.
Sedentary behaviour | 6 months (all groups)
  Sedentary behaviour will be evaluated using a Screen Time Questionnaire (STQ). The total screen hours will ba obtained by measuring: hours of daily TV, weekend TV, daily Computer, weekend computer, daily videogames, weekend videogames, daily free internet, weekend free internet, daily study internet, weekend study internet, and weekend study.
Sleep habits | Baseline (all groups)
  Sleep habits will be evaluated using the Pediatric Sleep Questionnaire (PSQ) (no units).
Sleep habits | 6 months (all groups)
  Sleep habits will be evaluated using the Pediatric Sleep Questionnaire (PSQ) (no units).
Eating disorders - SCOFF Questionnaire | Baseline (all groups)
  SCOFF questionnaire for the screening of eating disorders in primary care. Units: SCOFF score. Score>2, positive screening
Eating disorders - SCOFF Questionnaire | 6 months (all groups)
  SCOFF questionnaire for the screening of eating disorders in primary care. Units: SCOFF score. Score>2, positive screening
Eating disorders- DEBQ Questionnaire | Baseline (all groups)
  Dutch Eating Behavior Questionnaire for Children (DEBQ-C). Units: DEBQ score. The questionnaire measures three eating behaviors: emotional, external and restrained.
Eating disorders- DEBQ Questionnaire | 6 months (all groups)
  Dutch Eating Behavior Questionnaire for Children (DEBQ-C). Units: DEBQ score. The questionnaire measures three eating behaviors: emotional, external and restrained.
Plasma glucose | Baseline (all groups)
  Gucose (mg/dL)
Plasma glucose | 6 months (all groups)
  Gucose (mg/dL)
Plasma insulin | Baseline (all groups)
  Insulin (mg/dL)
Plasma insulin | 6 months (all groups)
  Insulin (mg/dL)
Plasma triglycerides (TG) | Baseline (all groups)
  TG (mg/dL)
Plasma triglycerides (TG) | 6 months (all groups)
  TG (mg/dL)
Plasma total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) | Baseline (all groups)
  Total cholesterol, HDL-C and LDL-C (mg/dL)
Plasma total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) | 6 months (all groups)
  Total cholesterol, HDL-C and LDL-C (mg/dL)
Plasma uric acid | Baseline (all groups)
  Uric acid (mg/dL)
Plasma uric acid | 6 months (all groups)
  Uric acid (mg/dL)
Plasma creatinine | Baseline (all groups)
  Creatinine (mg/dL)
Plasma creatinine | 6 months (all groups)
  Creatinine (mg/dL)
Insulin resistance | Baseline (all groups)
  Insulin resistance will be assessed by the homeostatic model assessment (HOMA) index
Insulin resistance | 6 months (all groups)
  Insulin resistance will be assessed by the homeostatic model assessment (HOMA) index
Analysis of additional circulating metabolites | Baseline (all groups)
  Metabolites (including myokines and adipokines) will be assessed using commercial enzyme-linked immunosorbent assays (ELISA)
Analysis of additional circulating metabolites | 6 months (all groups)
  Metabolites (including myokines and adipokines) will be assessed using commercial enzyme-linked immunosorbent assays (ELISA)
Transcriptome analysis | Baseline (all groups)
  Transcriptome analysis will be performed with RNA Sequencing (RNA-Seq) using next-generation sequencing platforms in peripheral blood cells (PBC)
Transcriptome analysis | 6 months (all groups)
  Transcriptome analysis will be performed with RNA Sequencing (RNA-Seq) using next-generation sequencing platforms in peripheral blood cells (PBC)
Circulating miRNA | Baseline (all groups)
  Circulating miRNA will be analysed using miRCURY LNA miRNA miRNome PCR Panels (Qiagen)
Circulating miRNA | 6 months(all groups)
  Circulating miRNA will be analysed using miRCURY LNA miRNA miRNome PCR Panels (Qiagen)
Evaluation of metabolomics and lipidomics | Baseline (all groups)
  Untargeted and targeted metabolomics and lipidomics will also be performed in plasma using liquid chromatography - mass spectrometry-based (LC-MS) methods.
Evaluation of metabolomics and lipidomics | 6 months (all groups)
  Untargeted and targeted metabolomics and lipidomics will also be performed in plasma using liquid chromatography - mass spectrometry-based (LC-MS) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Catalina Picó, Prof., Principal Investigator — Fundació d'investigació Sanitària de les Illes Balears; Empar Lurbe, Prof., Principal Investigator — General University Hospital Consortium of Valencia
Locations (1):
- General University Hospital Consortium of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data sets will be available on a restricted basis during the project. When the project is complete, the data will be freely accessible after an embargo period. In any case, personal data will not be freely accessible.
Time Frame: The data will be available directly within the project Consortium. Thus, access to these data will be approved by the project coordination board.
Access Criteria: The raw data will be recorded and deposited in an open repository, the "ELIXIR Core Data Resources". A two-year embargo period will apply to ensure a period of exclusive use of the data for INTEGRactiv Consortium partners.

REFERENCES:
- [Derived] Pico C, Lurbe E, Keijer J, Kopecky J, Landrier JF, Alvarez-Pitti J, Martin JC, Oliver P, Palou A, Palou M, Zouhar P, Ribot J, Rodriguez AM, Sanchez J, Serra F, Bonet ML. Study protocol: Identification and validation of integrative biomarkers of physical activity level and health in children and adolescents (INTEGRActiv). Front Pediatr. 2023 Sep 12;11:1250731. doi: 10.3389/fped.2023.1250731. eCollection 2023. PMID 37772038